CLINICAL TRIAL: NCT01016912
Title: A Phase 2a Study of BMS-790052 in Combination With Peginterferon Alfa-2b (PegIntron®) and Ribavirin (Rebetol®) in Japanese Subjects With Genotype 1 Chronic Hepatitis C Virus (HCV) Infection
Brief Title: Safety and Efficacy of Daclatasvir (BMS-790052) Plus Standard of Care (Pegylated-interferon Alpha-2b and Ribavirin) in Japanese Patients
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AI444-021
Record Dates: First submitted 2009-11-19; First posted 2009-11-20 (Estimated); Results first posted 2015-10-12 (Estimated); Last update posted 2015-10-12 (Estimated); Status verified 2015-09

CONDITIONS: Hepatitis C Infection
MeSH Terms: conditions — Hepatitis C | interventions — daclatasvir; peginterferon alfa-2b; Ribavirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (5):
- Arm A (BMS-790052, plus Peginterferon alfa-2b, Ribavirin) (Experimental): Treatment Naive
  Interventions: Drug: BMS-790052; Drug: Peginterferon alfa-2b; Drug: Ribavirin
- Arm B (BMS-790052, plus Peginterferon alfa-2b, Ribavirin) (Experimental): Treatment Naive
  Interventions: Drug: BMS-790052; Drug: Peginterferon alfa-2b; Drug: Ribavirin
- Arm C (Placebo, plus Peginterferon alfa-2b, Ribavirin) (Placebo Comparator): Treatment Naive
  Interventions: Drug: Placebo; Drug: Peginterferon alfa-2b; Drug: Ribavirin
- Arm D (BMS-790052, plus peginterferon alfa-2b, Ribavirin) (Experimental): Non-Responder
  Interventions: Drug: BMS-790052; Drug: Peginterferon alfa-2b; Drug: Ribavirin
- Arm E (BMS-790052, plus Peginterferon alfa-2b, Ribavirin) (Experimental): Non-Responder
  Interventions: Drug: BMS-790052; Drug: Peginterferon alfa-2b; Drug: Ribavirin

INTERVENTIONS:
Drug: BMS-790052 — Tablets, Oral, 10 mg, daily, 24-48 weeks
  Arms: Arm A (BMS-790052, plus Peginterferon alfa-2b, Ribavirin); Arm D (BMS-790052, plus peginterferon alfa-2b, Ribavirin)
Drug: BMS-790052 — Tablets, Oral, 60 mg, daily, 24-48 weeks
  Arms: Arm B (BMS-790052, plus Peginterferon alfa-2b, Ribavirin); Arm E (BMS-790052, plus Peginterferon alfa-2b, Ribavirin)
Drug: Placebo — Tablets, Oral, 0 mg, daily, 48 weeks
  Arms: Arm C (Placebo, plus Peginterferon alfa-2b, Ribavirin)
Drug: Peginterferon alfa-2b — Syringe, Subcutaneous, 180µg, weekly, 24-48 weeks
  Other Names: PegIntron®
Drug: Ribavirin — Capsules, Oral, 600 to 1000 mg based on weight, daily, 24-48 weeks
  Other Names: Rebetol®

SUMMARY:
The purpose of this study is to identify at least 1 dose of daclatasvir that is safe, well tolerated, and efficacious when combined with peginterferon-alfa and ribavirin for the treatment of hepatitis C virus genotype 1 in chronically infected patients who are treatment-naïve and nonresponsive to the standard of care

ELIGIBILITY:
Key Inclusion Criteria:

* Patients chronically infected with hepatitis C virus (HCV) genotype 1
* HCV RNA viral load ≥10*5* IU/mL at screening
* Naïve or nonresponsive to the current standard of care

Key Exclusion Criteria:

* Cirrhosis
* Hepatocellular carcinoma
* Coinfection with hepatitis B virus, HIV-1 or HIV-2

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2009-12; Primary Completion 2010-09 (Actual); Study Completion 2010-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (6):
- Japan (6):
  - Local Institution, Hiroshima, Hiroshima
  - Local Institution, Sapporo, Hokkaido
  - Local Institution, Kawasaki-Shi, Kanagawa
  - Local Institution, Suita-Shi, Osaka
  - Local Institution, Iruma-Gun, Saitama
  - Local Institution, Minato-Ku, Tokyo

REFERENCES:
- [Derived] Murakami E, Imamura M, Hayes CN, Abe H, Hiraga N, Honda Y, Ono A, Kosaka K, Kawaoka T, Tsuge M, Aikata H, Takahashi S, Miki D, Ochi H, Matsui H, Kanai A, Inaba T, McPhee F, Chayama K. Ultradeep sequencing study of chronic hepatitis C virus genotype 1 infection in patients treated with daclatasvir, peginterferon, and ribavirin. Antimicrob Agents Chemother. 2014;58(4):2105-12. doi: 10.1128/AAC.02068-13. Epub 2014 Jan 27. PMID 24468783
- See also: Investigator Inquiry form — http://www.bms.com/clinical_trials/Pages/Investigator_Inquiry_form.aspx

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 sites in Japan.
Pre-assignment Details: A total of 51 participants were enrolled, of which 45 were randomized to receive treatment and 6 were discontinued for no longer meeting study criteria.
Groups:
- Placebo + pegIFNα + Ribavirin (Treatment-naive): Participants received a matching placebo of daclatasvir tablet, once daily coadministered with ribavirin, twice daily, and peginterferon alpha (pegIFNα) injection, once weekly. Treatment-naive participants were those who had never been exposed to any hepatitis C virus (HCV) therapy with interferon IFNα-containing regimens, including pegIFNα/ribavirin.
- Daclatasvir 10- mg + pegIFNα + Ribavirin (Treatment-naive): Participants received 10 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and peginterferon alpha-2b (pegIFNα) injection, once weekly. Treatment-naive participants were those who had never been exposed to any hepatitis C virus (HCV) therapy with interferon IFNα-containing regimens, including pegIFNα/ribavirin.
- Daclatasvir 60- mg + pegIFNα + Ribavirin (Treatment-naive): Participants received 60 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection, once weekly. Treatment-naive participants were those who had never been exposed to any HCV therapy with interferon IFNα-containing regimens, including pegIFNα/ribavirin.
- Daclatasvir 10- mg + pegIFNα+ Ribavirin (Nonresponders): Participants received 10 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection once weekly. Nonresponders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care, pegIFNα/ribavirin.
- Daclatasvir 60- mg + pegIFNα + Ribavirin (Nonresponders): Participants received 60 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection once weekly. Nonresponders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care pegIFNα/ribavirin.
Period: End of Treatment Period
Arm/Group | Placebo + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10- mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 60- mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10- mg + pegIFNα+ Ribavirin (Nonresponders) | Daclatasvir 60- mg + pegIFNα + Ribavirin (Nonresponders)
Started | 8 | 9 | 10 | 9 | 9
Received Treatment | 8 | 9 | 10 | 9 | 9
Completed | 8 | 6 | 9 | 5 | 5
Not Completed | 0 | 3 | 1 | 4 | 4
Not completed — Lack of Efficacy | 0 | 1 | 0 | 4 | 4
Not completed — Adverse Event | 0 | 1 | 1 | 0 | 0
Not completed — Completed double-blind period only | 0 | 1 | 0 | 0 | 0
Period: Follow-up Period
Arm/Group | Placebo + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10- mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 60- mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10- mg + pegIFNα+ Ribavirin (Nonresponders) | Daclatasvir 60- mg + pegIFNα + Ribavirin (Nonresponders)
Started | 8 | 9 (Those who completed period 1 or with detectable hepatitis C virus RNA, despite length of treatment) | 10 (Those who completed period 1 or with detectable hepatitis C virus RNA, despite length of treatment) | 9 (Those who completed period 1 or with detectable hepatitis C virus RNA, despite length of treatment) | 9 (Those who completed period 1 or with detectable hepatitis C virus RNA, despite length of treatment)
Completed | 8 | 9 | 9 | 8 | 9
Not Completed | 0 | 0 | 1 | 1 | 0
Not completed — Other reason | 0 | 0 | 1 | 1 | 0

BASELINE CHARACTERISTICS:
Population: All treated participants who received at least 1 dose of study therapy.
Groups:
- Placebo + pegIFNα + Ribavirin (Treatment-naive): Participants received a matching placebo of daclatasvir tablet, once daily coadministered with ribavirin, twice daily, and peginterferon alpha-2b (pegIFNα) injection, once weekly. Treatment-naive participants were those who had never been exposed to any hepatitis C virus (HCV) therapy with interferon IFNα-containing regimens, including pegIFNα/ribavirin.
- Daclatasvir 10- mg + pegIFNα- + Ribavirin (Treatment-naive): Participants received 10 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection, once weekly. Treatment-naive participants were those who had never been exposed to any HCV therapy with interferon IFNα-containing regimens, including pegIFNα/ribavirin.
- Daclatasvir 10- mg + pegIFNα + Ribavirin (Nonresponders): Participants received 10 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection once weekly. Nonresponders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care, pegIFNα/ribavirin.
- Total: Total of all reporting groups
Arm/Group | Placebo + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10- mg + pegIFNα- + Ribavirin (Treatment-naive) | Daclatasvir 60- mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10- mg + pegIFNα + Ribavirin (Nonresponders) | Daclatasvir 60- mg + pegIFNα + Ribavirin (Nonresponders) | Total
Number analyzed (Participants) | 8 | 9 | 10 | 9 | 9 | 45
Age, Continuous [Mean (Standard Deviation); unit: years] | 52.6 (8.78) | 49.1 (15.09) | 53.2 (9.96) | 57.4 (6.11) | 58.8 (9.46) | 54.2 (10.46)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 7 | 4 | 6 | 6 | 27
  Male | 4 | 2 | 6 | 3 | 3 | 18

OUTCOME MEASURES:

1. Other Pre Specified Outcome: Number of Participants With Serious Adverse Events (SAEs), Discontinuations Due to Adverse Events (AEs), Treatment-related AEs, and Death as Outcome
Description: AE was defined as any new unfavorable symptom, sign, or disease or worsening of a preexisting condition that does not has a causal relationship with treatment. SAE was defined as a medical event that at any dose resulted in death, persistent or significant disability/incapacity, or drug dependency/abuse; was life-threatening, an important medical event, or a congenital anomaly/birth defect; or required or prolonged hospitalization. Treatment-related AE was defined as an AE that had certain, probable, possible, or unknown relationship to study drug.
Time Frame: From baseline to 30 days after last dose of study drug
Population: All participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Groups:
- Placebo + pegIFNα + Ribavirin (Treatment-naive): Participants received a matching placebo of daclatasvir tablet, once daily coadministered with ribavirin, twice daily, and peginterferon alpha(pegIFNα) injection, once weekly. Treatment-naive participants were those who had never been exposed to any hepatitis C virus (HCV) therapy with interferon IFNα-containing regimens, including pegIFNα/ribavirin.
- Daclatasvir 10- mg+ pegIFNα + Ribavirin (Nonresponders): Participants received 10 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection once weekly. Nonresponders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care pegIFNα/ribavirin.
- Daclatasvir 60- mg + pegIFNα- + Ribavirin (Nonresponders): Participants received 60 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection once weekly. Nonresponders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care pegIFNα/ribavirin.
Arm/Group | Placebo + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10- mg + pegIFNα- + Ribavirin (Treatment-naive) | Daclatasvir 60- mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10- mg+ pegIFNα + Ribavirin (Nonresponders) | Daclatasvir 60- mg + pegIFNα- + Ribavirin (Nonresponders)
Number analyzed (Participants) | 8 | 9 | 10 | 9 | 9
participants
  SAEs | 0 | 0 | 0 | 1 | 0
  Discontinuation due to AEs | 0 | 1 | 1 | 0 | 0
  Treatment-related AEs | 8 | 9 | 10 | 9 | 9
  Death | 0 | 0 | 0 | 0 | 0

2. Other Pre Specified Outcome: Number of Participants With Grade 3 to 4 Abnormalities on Laboratory Test Results
Description: Clinically significant marked abnormalities in laboratory test results graded by the Division of AIDS grading table, 2004. Hemoglobin: Grade 3= <7.0 to 8.9 g/dL, Grade 4= <7.0 g/dL. Lymphocytes: Grade 3= 350-499 cells/mm^3, Grade 4= <350 cells/mm^3. Neutrophils: Grade 3= 500-999 cells/mm^3, Grade 4= <500 cells/mm^3. White blood cells (WBC): Grade 3= 1000-1499 cells/mm^3, Grade 4= <1000 cells/mm^3. Alanine aminotransferase (ALT): Grade 3= 5.1-10*upper limit of normal (ULN), Grade 4= >10.0*ULN. Aspartate aminotransferase (AST): Grade 3= 5.1-10*ULN, Grade 4= >10.0*ULN. Total bilirubin: Grade 3= 2.6-5*ULN, Grade 4= >5.0*ULN.
Time Frame: From baseline to 30 days after last dose of study drug
Population: All participants who received at least 1 dose of study therapy.
Measure: Number; unit: participants
Groups:
- Daclatasvir 10- mg + pegIFNα + Ribavirin (Treatment-naive): Participants received 10 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection, once weekly. Treatment-naive participants were those who had never been exposed to any HCV therapy with interferon IFNα-containing regimens, including pegIFNα/ribavirin..
- Daclatasvir 60- mg + pegIFNα- + Ribavirin (Treatment-naive): Participants received 60 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection, once weekly. Treatment-naive participants were those who had never been exposed to any HCV therapy with interferon IFNα-containing regimens, including pegIFNα/ribavirin.
- Daclatasvir 60- mg + pegIFNα- + Ribavirin (Nonresponders): Participants received 60 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection once weekly. Nonresponders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care, pegIFNα/ribavirin.
Arm/Group | Placebo + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10- mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 60- mg + pegIFNα- + Ribavirin (Treatment-naive) | Daclatasvir 10- mg + pegIFNα + Ribavirin (Nonresponders) | Daclatasvir 60- mg + pegIFNα- + Ribavirin (Nonresponders)
Number analyzed (Participants) | 8 | 9 | 10 | 9 | 9
participants
  Hemoglobin | 1 | 0 | 1 | 3 | 0
  Lymphocytes | 2 | 2 | 3 | 3 | 2
  Neutrophils | 2 | 4 | 2 | 2 | 0
  WBC | 1 | 1 | 0 | 2 | 0
  ALT | 0 | 1 | 0 | 0 | 1
  AST | 0 | 1 | 0 | 0 | 1
  Total bilirubin | 0 | 1 | 0 | 0 | 0

3. Primary Outcome: Percentage of Participants With Extended Rapid Virologic Response (eRVR)
Description: eRVR was defined as undetectable hepatitis C virus (HCV) RNA (ie, HCV RNA <15 IU/mL, the lower limit of detection, target not detected) at both Weeks 4 and 12. HCV RNA levels were measured by Tobas TaqMan HCV Auto from the central laboratory.
Time Frame: At Weeks 4 and 12 on treatment
Population: All participants who received at least 1 dose of study therapy.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir 60- mg + pegIFNα + Ribavirin (Treatment Naive): Participants received 60 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection, once weekly. Treatment-naive participants were those who had never been exposed to any HCV therapy with interferon IFNα-containing regimens, including pegIFNα/ribavirin.
- Daclatasvir 10- mg + pegINFα + Ribavirin (Nonresponders): Participants received 10 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection once weekly. Nonresponders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care, pegIFNα/ribavirin.
Arm/Group | Placebo + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10- mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 60- mg + pegIFNα + Ribavirin (Treatment Naive) | Daclatasvir 10- mg + pegINFα + Ribavirin (Nonresponders) | Daclatasvir 60- mg + pegIFNα + Ribavirin (Nonresponders)
Number analyzed (Participants) | 8 | 9 | 10 | 9 | 9
percentage of participants | 0 [0.0 to 25.0] | 66.7 [40.1 to 87.1] | 80.0 [55.0 to 94.5] | 55.6 [30.1 to 79.0] | 22.2 [6.1 to 49.0]

4. Secondary Outcome: Percentage of Participants With Rapid Virologic Response (RVR)
Description: RVR was defined as undetectable hepatitis C virus (HCV) RNA (ie, HCV RNA <15 IU/mL, the lower limit of detection, target not detected) at Week 4. HCV RNA levels were measured by CobasTaqMan HCV Auto from the central laboratory .
Time Frame: At Week 4 on treatment
Population: All participants who received at least 1 dose of study therapy.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir 10 mg + pegIFNα + Ribavirin (Treatment-naive): Participants received 10 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection, once weekly. Treatment-naive participants were those who had never been exposed to any HCV therapy with interferon IFNα-containing regimens, including pegIFNα/ribavirin.
- Daclatasvir 60 mg + pegIFNα + Ribavirin (Treatment-naive): Participants received 60 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection, once weekly. Treatment-naive participants were those who had never been exposed to any HCV therapy with interferon IFNα-containing regimens, including pegIFNα/ribavirin.
- Daclatasvir 10 mg + pegIFNα + Ribavirin (Nonresponders): Participants received 10 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection once weekly. Nonresponders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care, pegIFNα/ribavirin..
- Daclatasvir 60 mg + pegIFNα + Ribavirin (Nonresponders): Participants received 60 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection once weekly. Nonresponders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care pegIFNα/ribavirin.
Arm/Group | Placebo + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10 mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 60 mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10 mg + pegIFNα + Ribavirin (Nonresponders) | Daclatasvir 60 mg + pegIFNα + Ribavirin (Nonresponders)
Number analyzed (Participants) | 8 | 9 | 10 | 9 | 9
percentage of participants | 0 [0.0 to 25.0] | 77.8 [51.0 to 93.9] | 80.0 [55.0 to 94.5] | 55.6 [30.1 to 79.0] | 33.3 [12.9 to 59.9]

5. Secondary Outcome: Percentage of Participants With Complete Early Virologic Response (cEVR)
Description: cEVR was defined as undetectable hepatitis C virus (HCV) RNA (ie, HCV RNA <15 IU/mL, the lower limit of detection, target not detected) at Week 12 on treatment. HCV RNA levels were measured by Cobas TaqMan HCV Auto from the central laboratory
Time Frame: At Week 12 on treatment
Population: All participants who received at least 1 dose of study therapy.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir 10 mg + pegIFNα + Ribavirin (Nonreponders): Participants received 10 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection once weekly. Nonresponders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care, pegIFNα/ribavirin.
Arm/Group | Placebo + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10 mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 60 mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10 mg + pegIFNα + Ribavirin (Nonreponders) | Daclatasvir 60 mg + pegIFNα + Ribavirin (Nonresponders)
Number analyzed (Participants) | 8 | 9 | 10 | 9 | 9
percentage of participants | 62.5 [34.5 to 85.3] | 77.8 [51.0 to 93.9] | 100.0 [79.4 to 100.0] | 55.6 [30.1 to 79.0] | 55.6 [30.1 to 79.0]

6. Secondary Outcome: Percentage of Participants With a Sustained Virologic Response (SVR) at Weeks 4, 12, and 24
Description: SVR at follow-up Week 4 (SVR4), follow-up Week 12 (SVR12), and follow-up Week 24 (SVR24) is defined as undetectable hepatitis C virus (HCV) RNA (ie, HCV RNA <15 IU/mL, the lower limit of detection, target not detected) at each of these timepoints. HCV RNA levels were measured by Cobas TaqMan HCV Auto from the central laboratory .
Time Frame: Follow-up Weeks 4, 12, and 24
Population: All participants who received at least 1 dose of study therapy.
Measure: Number (80% Confidence Interval); unit: percentage of participants
Groups:
- Daclatasvir 60 mg + pegIFNα + Ribavirin (Nonresponders): Participants received 60 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection once weekly. Nonresponders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care, pegIFNα/ribavirin
Arm/Group | Placebo + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10 mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 60 mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10 mg + pegIFNα + Ribavirin (Nonresponders) | Daclatasvir 60 mg + pegIFNα + Ribavirin (Nonresponders)
Number analyzed (Participants) | 8 | 9 | 10 | 9 | 9
percentage of participants
  SVR4: Follow-up Week 4 | 75.0 [46.2 to 93.1] | 66.7 [40.1 to 87.1] | 90.0 [66.3 to 99.0] | 22.2 [6.1 to 49.0] | 33.3 [12.9 to 59.9]
  SVR12: Follow-up Week 12 | 62.5 [34.5 to 85.3] | 66.7 [40.1 to 87.1] | 90.0 [66.3 to 99.0] | 22.2 [6.1 to 49.0] | 33.3 [12.9 to 59.9]
  SVR24: Follow-up Week 24 | 62.5 [34.5 to 85.3] | 66.7 [40.1 to 87.1] | 90.0 [66.3 to 99.0] | 22.2 [6.1 to 49.0] | 33.3 [12.9 to 59.9]

7. Secondary Outcome: Percentage of Participants With Virologic Failure
Description: Virologic failure is defined by the following 6 categories: 1.Virologic breakthrough, defined as confirmed >1 log10 increase in hepatitis C virus (HCV) RNA over nadir or confirmed HCV RNA ≥limit of quantitation (LOQ) after confirmed undetectable HCV RNA while on treatment. 2. <1 log10 decrease in HCV RNA from baseline at Week 4 of treatment. 3. Failure to achieve early virologic response, defined as <2 log10 decrease in HCV RNA from baseline at Week 12 of treatment. 4. Detectable HCV RNA at Week 12, and HCV RNA ≥LOQ at Week 24 of treatment. 5. Detectable HCV RNA at end of treatment (including early discontinuation). 6 Relapse, defined as detectable HCV RNA during follow-up after undetectable HCV RNA levels at end of treatment.
Time Frame: From on-treatment Week 1 to Follow-up Week 24
Population: All participants who received at least 1 dose of study therapy.
Measure: Number; unit: percentage of participants
Groups:
- Daclatasvir 60 mg + Peg-IFNα + Ribavirin (Treatment-naive): received 60 mg of daclatasvir, once daily, coadministered with ribavirin, twice daily, and pegIFNα injection, once weekly. Treatment-naive participants were those who had never been exposed to any HCV therapy with interferon IFNα-containing regimens, including pegIFNα/ribavirin.
Arm/Group | Placebo + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 10 mg + pegIFNα + Ribavirin (Treatment-naive) | Daclatasvir 60 mg + Peg-IFNα + Ribavirin (Treatment-naive) | Daclatasvir 10 mg + pegIFNα + Ribavirin (Nonresponders) | Daclatasvir 60 mg + pegIFNα + Ribavirin (Nonresponders)
Number analyzed (Participants) | 8 | 9 | 10 | 9 | 9
percentage of participants
  Virologic failure | 37.5 | 33.3 | 10.0 | 77.8 | 66.7
  Virologic breakthrough | 12.5 | 11.1 | 0.0 | 44.4 | 44.4
  Relapse | 25.0 | 11.1 | 10.0 | 33.3 | 22.2

ADVERSE EVENTS:
Time Frame: From baseline up to 30 days after last dose of study drug
Groups:
- Placebo+pegIFNα +Ribavirin (Treatment Naive): Participants received a matching placebo of daclatasvir tablet, orally, once daily (OD) with peginterferon alpha-2a (pegIFNα) subcutaneously once weekly and ribavirin orally, twice daily (BID). Treatment naive participants were those who had never been exposed to any Hepatitis C Virus (HCV) therapy with interferon IFNα containing regimens including pegIFNα-2b/ribavirin.
- Daclatasvir 10- mg+pegIFNα+Ribavirin (Treatment Naive): Participants received 10 mg of daclatasvir OD coadministered with pegIFNα subcutaneously once weekly and ribavirin orally BID. Treatment naive participants were defined as those who had never been exposed to any HCV therapy with IFNα containing regimens including pegIFNα-2b/ribavirin.
- Daclatasvir 60- mg+pegIFNα+Ribavirin (Treatment Naive): Participants received 60 mg of daclatasvir OD in coadministration with pegIFNα administered subcutaneously once weekly and ribavirin administered orally BID. Treatment naive participants were defined as those who had never been exposed to any HCV therapy with IFNα containing regimens including pegIFNα-2b/ribavirin.
- Daclatasvir 10- mg+pegIFNα+Ribavirin (Non--Responders): Participants received 10 mg of daclatasvir OD coadministered with pegIFNα subcutaneously once weekly and ribavirin orally BID. Non-responders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care pegIFNα-2b/ribavirin.
- Daclatasvir 60- mg+pegIFNα+Ribavirin (Non--Responders): Participants received 60 mg of daclatasvir OD in coadministration with pegIFNα administered subcutaneously once weekly and ribavirin administered orally BID. Non-responders were participants who had never attained undetectable HCV RNA levels, after at least 12 weeks of the current standard of care pegIFNα-2b/ribavirin.
Arm/Group | Placebo+pegIFNα +Ribavirin (Treatment Naive) | Daclatasvir 10- mg+pegIFNα+Ribavirin (Treatment Naive) | Daclatasvir 60- mg+pegIFNα+Ribavirin (Treatment Naive) | Daclatasvir 10- mg+pegIFNα+Ribavirin (Non--Responders) | Daclatasvir 60- mg+pegIFNα+Ribavirin (Non--Responders)
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/9 | 0/10 | 1/9 | 0/9
Other Adverse Events (participants affected / at risk) | 8/8 | 9/9 | 10/10 | 9/9 | 9/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+pegIFNα +Ribavirin (Treatment Naive) (N=8) | Daclatasvir 10- mg+pegIFNα+Ribavirin (Treatment Naive) (N=9) | Daclatasvir 60- mg+pegIFNα+Ribavirin (Treatment Naive) (N=10) | Daclatasvir 10- mg+pegIFNα+Ribavirin (Non--Responders) (N=9) | Daclatasvir 60- mg+pegIFNα+Ribavirin (Non--Responders) (N=9)
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo+pegIFNα +Ribavirin (Treatment Naive) (N=8) | Daclatasvir 10- mg+pegIFNα+Ribavirin (Treatment Naive) (N=9) | Daclatasvir 60- mg+pegIFNα+Ribavirin (Treatment Naive) (N=10) | Daclatasvir 10- mg+pegIFNα+Ribavirin (Non--Responders) (N=9) | Daclatasvir 60- mg+pegIFNα+Ribavirin (Non--Responders) (N=9)
Amenorrhoea (Reproductive system and breast disorders) | 0 | 0 | 0 | 1 | 0
Blood thyroid stimulating hormone increased (Investigations) | 2 | 0 | 0 | 0 | 0
Dermatitis acneiform (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dermatitis atopic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Dizziness (Nervous system disorders) | 0 | 0 | 1 | 2 | 1
Dysgeusia (Nervous system disorders) | 0 | 0 | 3 | 3 | 0
Eye pain (Eye disorders) | 0 | 0 | 0 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0 | 1
Fatigue (General disorders) | 3 | 0 | 3 | 3 | 1
Feeling abnormal (General disorders) | 0 | 0 | 1 | 0 | 0
Gastroenteritis (Infections and infestations) | 0 | 0 | 0 | 1 | 0
Hypothyroidism (Endocrine disorders) | 0 | 0 | 0 | 1 | 1
Injection site rash (General disorders) | 0 | 0 | 1 | 0 | 0
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 0 | 1 | 1 | 0 | 0
Neutropenia (Blood and lymphatic system disorders) | 2 | 4 | 2 | 2 | 0
Retinal tear (Eye disorders) | 1 | 0 | 0 | 0 | 0
Retinopathy (Eye disorders) | 1 | 0 | 0 | 0 | 0
Vertigo (Ear and labyrinth disorders) | 0 | 0 | 0 | 0 | 1
Anxiety disorder (Psychiatric disorders) | 0 | 0 | 0 | 0 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 0 | 0
Depressed mood (Psychiatric disorders) | 1 | 0 | 0 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 1 | 3 | 4 | 3 | 1
Dry mouth (Gastrointestinal disorders) | 0 | 0 | 1 | 1 | 0
Epigastric discomfort (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 0 | 0
Folliculitis (Infections and infestations) | 1 | 0 | 0 | 0 | 0
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Lymphopenia (Blood and lymphatic system disorders) | 2 | 2 | 3 | 3 | 2
Nail disorder (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Nasopharyngitis (Infections and infestations) | 2 | 5 | 3 | 0 | 2
Neuropathy peripheral (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Prurigo (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 0 | 1
Temporomandibular joint syndrome (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Thermal burn (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
Ventricular extrasystoles (Cardiac disorders) | 0 | 1 | 0 | 0 | 0
Vessel puncture site pain (General disorders) | 0 | 0 | 0 | 1 | 0
Weight decreased (Investigations) | 3 | 0 | 0 | 1 | 1
Ear pain (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Injection site reaction (General disorders) | 1 | 1 | 2 | 2 | 1
Laryngeal inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Nasal congestion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 0 | 0 | 0
Alanine aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 0 | 0 | 0
Blepharitis (Eye disorders) | 0 | 1 | 1 | 0 | 0
Blood triglycerides increased (Investigations) | 0 | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 0 | 0
Carpal tunnel syndrome (Nervous system disorders) | 0 | 1 | 0 | 0 | 0
Conjunctivitis (Eye disorders) | 0 | 1 | 0 | 0 | 0
Dyspepsia (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Dyspnoea exertional (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1 | 0
Migraine (Nervous system disorders) | 0 | 0 | 2 | 0 | 0
Neck mass (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal discomfort (Respiratory, thoracic and mediastinal disorders) | 1 | 1 | 0 | 0 | 0
Poor quality sleep (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Rash (Skin and subcutaneous tissue disorders) | 3 | 2 | 5 | 0 | 1
Retinal disorder (Eye disorders) | 1 | 0 | 0 | 0 | 0
Rhinitis allergic (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Abdominal distension (Gastrointestinal disorders) | 1 | 1 | 0 | 0 | 1
Anaemia (Blood and lymphatic system disorders) | 5 | 2 | 2 | 5 | 1
Arthropod sting (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0 | 0
Cheilitis (Gastrointestinal disorders) | 0 | 2 | 3 | 0 | 0
Chills (General disorders) | 0 | 0 | 2 | 1 | 0
Cystitis (Infections and infestations) | 0 | 0 | 0 | 2 | 2
Decreased appetite (Metabolism and nutrition disorders) | 1 | 3 | 3 | 5 | 2
Dizziness postural (Nervous system disorders) | 0 | 0 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 0 | 1
Influenza like illness (General disorders) | 0 | 1 | 1 | 2 | 1
Inner ear disorder (Ear and labyrinth disorders) | 0 | 0 | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Otitis externa (Infections and infestations) | 0 | 0 | 2 | 0 | 0
Pharyngitis (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Phosphenes (Eye disorders) | 1 | 0 | 0 | 0 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 3 | 3 | 2 | 1 | 5
Pruritus generalised (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 2 | 0
Urticaria (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0 | 1
Vessel puncture site reaction (General disorders) | 1 | 0 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 0 | 0 | 2 | 2 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 3 | 2 | 0 | 0 | 0
Atypical mycobacterial infection (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 3 | 1 | 1 | 1 | 2
Dental caries (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Injection site injury (General disorders) | 0 | 0 | 1 | 0 | 0
Leukopenia (Blood and lymphatic system disorders) | 1 | 1 | 0 | 2 | 0
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1 | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 1 | 1 | 2 | 0
Pyrexia (General disorders) | 5 | 8 | 9 | 6 | 8
Retinal haemorrhage (Eye disorders) | 0 | 0 | 0 | 1 | 0
Abdominal discomfort (Gastrointestinal disorders) | 1 | 2 | 3 | 1 | 1
Abdominal pain upper (Gastrointestinal disorders) | 0 | 2 | 0 | 0 | 1
Basedow's disease (Endocrine disorders) | 0 | 1 | 0 | 0 | 0
Dry eye (Eye disorders) | 1 | 0 | 0 | 0 | 1
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 0 | 0
Eczema asteatotic (Skin and subcutaneous tissue disorders) | 0 | 0 | 1 | 0 | 0
Enterocolitis (Gastrointestinal disorders) | 1 | 0 | 0 | 0 | 0
Injection site erythema (General disorders) | 1 | 2 | 0 | 0 | 0
Lip dry (Gastrointestinal disorders) | 1 | 0 | 1 | 0 | 0
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 1 | 0 | 0 | 0 | 0
Otitis media (Infections and infestations) | 0 | 0 | 1 | 0 | 0
Periodontitis (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 1
Retinal exudates (Eye disorders) | 0 | 0 | 1 | 0 | 0
Stomatitis (Gastrointestinal disorders) | 1 | 3 | 3 | 1 | 1
Syncope (Nervous system disorders) | 0 | 0 | 0 | 1 | 0
Tinnitus (Ear and labyrinth disorders) | 0 | 0 | 2 | 0 | 1
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0 | 0
Alopecia (Skin and subcutaneous tissue disorders) | 3 | 3 | 7 | 3 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 3 | 5 | 0
Blood phosphorus decreased (Investigations) | 0 | 0 | 1 | 0 | 0
Blood pressure increased (Investigations) | 1 | 0 | 0 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 2 | 0 | 0 | 0 | 1
Cough (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 2 | 0 | 1
Depression (Psychiatric disorders) | 0 | 0 | 1 | 0 | 0
Drug eruption (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Eczema (Skin and subcutaneous tissue disorders) | 1 | 1 | 2 | 2 | 0
Gingivitis (Gastrointestinal disorders) | 0 | 0 | 1 | 0 | 0
Headache (Nervous system disorders) | 5 | 6 | 4 | 5 | 3
Heat rash (Skin and subcutaneous tissue disorders) | 0 | 0 | 0 | 1 | 0
Injection site pruritus (General disorders) | 2 | 3 | 3 | 2 | 1
Insomnia (Psychiatric disorders) | 2 | 2 | 3 | 0 | 0
Lipase increased (Investigations) | 1 | 0 | 0 | 0 | 1
Malaise (General disorders) | 2 | 7 | 2 | 2 | 1
Myalgia (Musculoskeletal and connective tissue disorders) | 2 | 0 | 1 | 0 | 0
Oral herpes (Infections and infestations) | 0 | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0 | 0
Sputum retention (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0 | 0
Tachycardia (Cardiac disorders) | 0 | 0 | 0 | 0 | 1
Thrombocytopenia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 0 | 1
Vessel puncture site pruritus (General disorders) | 0 | 0 | 1 | 0 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Bristol Myers Squibb Co. agreements with investigators vary; constant is our right to embargo communications regarding trial results prior to public release for a period ≤60 days from submittal for review. We will not prohibit investigators from publishing, but will prohibit the disclosure of previously undisclosed confidential information other than study results, and request postponement of single center publications until after disclosure of the clinical trial's primary publication.